CLINICAL TRIAL: NCT04388449
Title: Multicenter Study on the Place of Intrathecal Analgesia to Improve the Quality of Life of Painful Cancer Patients: Development of a Grid for Analysing Life and Quality of Life
Brief Title: Place of Intrathecal Analgesia to Improve the Quality of Life of Painful Cancer Patients
Acronym: QUALITHEC01
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2019-18
Record Dates: First submitted 2020-04-09; First posted 2020-05-14 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-04

CONDITIONS: Injections, Spinal; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The intrathecal analgesia is a recommended technic to treat persistent pain in cancer patient but little used, whose the technical conditions require hospital multidisciplinary expertise and coordination associated to a link between city and hospital. The experience of patients who benefit of this technic in this situation of advanced cancer (loco-regional or metastatic) is little known. So far, it doesn't exist developed tools to know it.

In literature, 2 qualitative studies have been published on the quality of life with intrathecal analgesia. A study realised in 2009 with 6 Canadian patients (3 interview per patients) and nurses in palliative unit shows the positive impact on the quality of life of patients. Recently, a qualitative study has approached the question of the quality of life of patients who had an intrathecal analgesia with the point of view of nursing staff. The results confirm the improvement of quality of life and suggest an establishment more premature of technic in the care process.

Given the development of this technic in cancerology in France and more premature in the care process of patients, it seems interesting to know better the experience of patients with cancer and for who the pain is treated by this technic and the impact on the quality of life of these patients sometimes dependent of some expert centres. This study is done to answer to theses questions on the experience of patients and their close relations and the impact of the quality of life according to a qualitative approach. An independent psychologist of process care of patients will realised semi-directed before putting on the equipment allowing the administration of analgesic by intrathecal pathway, at 1 month, then 3 months to know the experience when the balance of the pain is generally reached (M1) and the impact in long-term (M3).

DETAILED DESCRIPTION:
The referent algologist informs the patient of the retained offer in the pain multidisciplinary consultation meeting. Following the consultation, the investigator sees the patient to explain the study and to verify all the inclusion and non-inclusion criteria, to give and explain the information note and to be sure of the non-opposition.

A psychologist comes in each centre to realise the semi-directed interviews before putting on the catheter, at 1 month and at 3 months after the establishment of this technic. The interview will be recorded with the agreement of the patient then totally transcribed. A double analysis will allow to extract the verbatim record and to construct the thematic tree with under-themes.

The same day of the interviews, 4 questionnaires will allow to evaluate to the 3 periods of measurement (before putting on the catheter, M1 et M3) : the mean pain of the past 24 hours by the BPI-SF (Brief Pain Inventory-short form) questionnaire, the anxiety and the depression by the HAD (Hospital Anxiety and Depression scale) questionnaire, the quality of life by the QLQ-C30 questionnaire, the catastrophism by the PCS (Pain Catastrophizing Scale) questionnaire.

The evaluation by the patient and the algologist of the global clinic improvement after the establishment of the analgesic treatment by intrathecal way will be realised at M1 and M3 with the help of the questionnaire P-GIC and C-GIC (Patient or Clinical- Global Impression of Change).

The study does not interfere with the treatment of the patient and his usual care. No biological exams or imagery will be realise in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is more than 18 years old with pain linked to the evolution of locoregional or distanced cancer justifying an analgesic treatment administrated by an intrathecal pathway with an implantable pump.
* Patient is able to answer to the questions during the semi-directed interview
* Patient has valid health insurance
* Having given written informed consent prior to any procedure related to the study

Exclusion Criteria:

* Patient under 18 years-old.
* Patient under guardianship or protection of vulnerable adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients having pain treated by analgesic administrated through an intrathecal way with an implantable pump will be included in this study.
  The inclusion of patients will be done with a consecutive way to avoid the selection bias. Each patient file will be presented to the pain multidisciplinary consultation meeting. It will have the validation of an antalgic treatment by an intrathecal way. The investigator will verify the inclusion and non-inclusion criteria to offer the study to all the corresponding patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the experience of patients who have an intrathecal analgesia treating nociceptive and/or neuropathic pain of cancerous origin in palliative phase. | 3 months
  The evaluation will done through a semi-structured interview by a psychologist. After the patient agreement, the interview is recorded so that can be fully transcribed. The recordings will be erased as soon as the transcription has been carried out completely anonymously. The data will be processed by a content analysis. It is a method of interpreting qualitative data which consists of an objective, exhaustive, methodical and if possible quantitative examination of communication material to classify its elements

SECONDARY OUTCOMES:
Evaluate the mean pain of the past 24 hours | 3 months
  The evaluation will be done through the Brief Pain Inventory-Short Form (BPI-SF) questionnaire. It is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning such as general activity, mood, walking ability, normal work including outside the home and housework, relations with other people, enjoyment of life, and sleep. This questionnaire is a 10 point scale (where 0 = no interference and 10 = interferes completely).
Evaluate the quality of life | 3 months
  The evaluation will be done through the QLQ-C30 questionnaire. It is a 30-item questionnaire composed by 4 dimensions (5 functional scales (cognitive, emotional, physical, role and social functioning), 3 symptom scales (fatigues, nausea/vomiting and pain) a global health status and 5 single items assessing additional symptoms (appetite loss, constipation, diarrhea, dyspnea and sleep disturbance)). The scales measures range score from 0 to 100. A high scale score represents a higher response level
Evaluate the pain catastrophizing | 3 months
  The evaluation will be done through the PCS (Pain Catastrophizing Scale) questionnaire. It is a 13-item questionnaire assessing rumination, magnification and helplessness about the pain. The PCS total score is computed by summing responses to all 13 items. PCS total scores range from 0 - 52. A high scale score represents a clinically relevant level of catastrophizing.
Evaluate the consistency of the feeling of the global clinic improvement of the patient | 3 months
  Using the PGIC (Patient Global Impression of Change) It is a 1-item questionnaire. The scale evaluates all aspects of patient health and assesses if there has been an improvement or decline in clinical status from 0 (much better) to 10 (much worse).
Evaluate the consistency or not of the feeling of the global clinic improvement of the clinician at M1 and M3. | 3 months
  Using the the CGIC (Clinical Global Impression of Change) It is is rated on a 7-point scale, with a severity of illness scale using a range of responses from 1 (very much improved) through to 7 ( very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Marie PECHARD, Study Director — Institut Curie
Locations (3):
- France (3):
  - Institut de Cancerologie de l'Ouest, Angers
  - INSERM U987 CHU A Paré - Institut Curie, Boulogne-Billancourt
  - Hopital Foch, Suresnes